CLINICAL TRIAL: NCT02324582
Title: Phase I Study of MK-3475 in Combination With BCG for Patients With High Risk Superficial Bladder Cancer
Brief Title: MK-3475/BCG in High Risk Superficial Bladder Cancer
Acronym: MARC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-SIUSOM-14-006
Record Dates: First submitted 2014-12-11; First posted 2014-12-24 (Estimated); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-04

CONDITIONS: Bladder Cancer
Keywords: Urinary Bladder Neoplasms; Mycobacterium bovis; Programmed Cell Death 1 Receptor; pembrolizumab
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous MK-3475/ Intravesical BCG (Experimental): 3 subjects will be treated at a dose of 100 mg MK-3475 at 100 mg every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses 12 subjects will be treated at a dose of 200 mg MK-3475 at 100 mg every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses
  Interventions: Drug: Intravenous MK-3475/ Intravesical BCG

INTERVENTIONS:
Drug: Intravenous MK-3475/ Intravesical BCG — 6 cycles (each cycle is 21 days) of pembrolizumab will be given over 9 weeks in combination with BCG. BCG treatment will begin on Day 1 of cycle 3 of pembrolizumab.
  Other Names: pembrolizumab

SUMMARY:
This is a single center Phase I safety and efficacy study of MK-3475 therapy used in combination with bladder infused BCG treatment for patients, 18 years or older, with high risk superficial bladder cancer (cancer not yet involving the muscle of the bladder wall) who have had removal of their bladder tumor. Patients will be enrolled to a single treatment group of a fixed dose of MK 3475 and BCG.

DETAILED DESCRIPTION:
Bladder cancer is the fifth most common cancer in the United States. This is a single center Phase I safety and efficacy study of MK-3475 therapy used in combination with bladder infused BCG treatment. The study will determine the safety of administering MK-3475 at a fixed dose every three weeks in conjunction with intravesicular BCG treatment in non-muscle invasive bladder cancer patients who had recurrence after two courses of induction (6 doses) intravesical therapy (two BCG courses, or one BCG course and one other approved intravesical therapies) administered within 12 months, or after one induction (6 doses) and one maintenance (3 doses) intravesical therapy (BCG). Subjects will have confirmation of bladder cancer non-invasive to the muscle. Approximately 20 subjects will be screened to treat 15 eligible subjects with high risk superficial bladder cancer who have had transurethral resection of their bladder tumor.

The rationale for the use of the indicated dose of TICE® BCG is based upon FDA approved and commercially provided package insert/ instructions for use of the product. BCG installation has been used to treat non-muscle-invasive bladder cancer for more than 30 years. It is one of the most successful biotherapies for cancer in use. Despite long clinical experience with BCG, the mechanism of its therapeutic effect is still under investigation.

The first 3 subjects will be treated at a dose of 100 mg MK-3475 to ensure safety for the combination. If no safety or efficacy issues are present, dosing will be escalated to 200 mg MK-3475 every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1.Willing and able to provide written informed consent/assent.

2.18 years of age.

3.Have pathologically documented high grade transitional cell superficial bladder cancer (Ta, T1) at time of restaging, or have pathologically documented high grade CIS of the bladder at time of initial resection for recurrent/persistent high risk transitional cell superficial bladder cancer.

4.Recurrent/persistent disease despite 2 Induction Intravesical Therapy Courses given within 12 months (with BCG being one of them), or despite one induction BCG treatment in addition to at least one maintenance course of BCG 5.Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion.

6.ECOG performance status of 0-2. 7.Demonstrate adequate organ function 8.Female subject of childbearing potential should have a negative urine or serum pregnancy.

9.Female subjects of childbearing potential should be willing to use 2 methods of birth control or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication 10.Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Currently has active or progressive metastatic disease.
2. Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Prior systemic chemotherapy, targeted small molecule therapy, or radiation therapy for bladder cancer.
6. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Known additional malignancy that is progressing or requires active treatment.
8. Active autoimmune disease that has required systemic treatment in past 2 years.
9. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
10. Active infection, including a concurrent febrile illness, requiring systemic therapy.
11. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 4 months after the last dose of trial treatment.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) including anti-CD40 and anti-OX40 antibodies.
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBs Ag reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Has known active tuberculosis. Subjects will not be specifically tested for the study; however, subjects that are tested within 28 days of beginning study or while on study and test positive with the PPD test before treatment should have active tuberculosis ruled out before therapy begins for their superficial bladder cancer.
18. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
19. Has an active urinary tract infection, gross hematuria, or known broken mucosal barrier of the bladder.
20. Less than 14 days post bladder biopsy, TUR, or traumatic catheterization.
21. Evidence of muscle invasive bladder cancer, or transitional cell carcinoma of the upper urinary tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Rao, MD, Principal Investigator — Southern Illinois University
Locations (3):
- United States (3):
  - Simmons Cancer Institute-SIU School of Medicine, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Henry Ford Health Systems, Detroit, Michigan

REFERENCES:
- [Derived] Jamil ML, Deebajah M, Sood A, Robinson K, Rao K, Sana S, Alanee S. Protocol for phase I study of pembrolizumab in combination with Bacillus Calmette-Guerin for patients with high-risk non-muscle invasive bladder cancer. BMJ Open. 2019 Jul 17;9(7):e028287. doi: 10.1136/bmjopen-2018-028287. PMID 31320352
- See also: Simmons Cancer Institute at Southern Illinois University School of Medicine — http://www.siumed.edu/cancer/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment for the study was open between 02 June 2015 through 10Oct 2019 in 2 urologic outpatient clinics.
Groups:
- Intravenous MK-3475-100 mg/ Intravesical BCG: 3 subjects will be treated at a dose of 100 mg MK-3475 at 100 mg every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses
  Intravenous MK-3475/ Intravesical BCG: 6 cycles (each cycle is 21 days) of pembrolizumab will be given over 9 weeks in combination with BCG. BCG treatment will begin on Day 1 of cycle 3 of pembrolizumab.
- Intravenous MK-3475-200 mg/ Intravesical BCG: Up to 12 Subjects will be treated at a dose of 200 mg MK-3475 at 100 mg every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses
Period: Overall Study
Arm/Group | Intravenous MK-3475-100 mg/ Intravesical BCG | Intravenous MK-3475-200 mg/ Intravesical BCG
Started | 3 (Enrollment open for dose of 100 mg MK-3475.) | 15 (Enrollment open for dose escalation to 200 mg MK-3475.)
Completed | 3 (Post treatment disease assessment for patient treated at 100 mg MK-3475 (pembrolizumab).) | 10 (Post treatment disease assessment for patient treated at 200 mg Mk-3475 (pembrolizumab).)
Not Completed | 0 | 5
Not completed — Screen Failures | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Intravenous MK-3475-100 mg/ Intravesical BCG: 3 subjects will be treated at a dose of 100 mg MK-3475 every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial (50 mg) intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses
  Intravenous MK-3475/ Intravesical BCG: 6 cycles (each cycle is 21 days) of pembrolizumab will be given over 19 weeks in combination with BCG. 6 cycles of BCG treatment will begin on Day 1 of cycle 3 of pembrolizumab.
- Intravenous MK-3475-200 mg/ Intravesical BCG: Up to 12 subjects will be treated at a dose of 200 mg MK-3475 every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial (50 mg) intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses
  Intravenous MK-3475/ Intravesical BCG: 6 cycles (each cycle is 21 days) of pembrolizumab will be given over 19 weeks in combination with BCG. 6 cycles of BCG treatment will begin on Day 1 of cycle 3 of pembrolizumab.
- Total: Total of all reporting groups
Arm/Group | Intravenous MK-3475-100 mg/ Intravesical BCG | Intravenous MK-3475-200 mg/ Intravesical BCG | Total
Number analyzed (Participants) | 3 | 10 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Full Range); unit: years] | 68 [55 to 75] | 70 [38 to 89] | 69 [38 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 3 | 8 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 9 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 10 | 13
Absence of tumor in the bladder following restaging resection. [Count of Participants; unit: Participants] — All subjects were required to have histologically confirmed high grade, non-muscle invasive bladder cancer at study entry and undergone restaging resection within 28 days of Day1 Week 1.
  Participants | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3, 4, and 5 Treatment Related Adverse Events
Description: Grade and quantity of treatment related adverse events. Due to the small sampling of subjects, no statistical analysis will be performed. Descriptive statistics in the form of counts calculated as percentages will be reported.
Time Frame: change from baseline to 23 weeks
Population: Thirteen patients were dosed (3 with 100mg MK3475 and 10 with 200 mg MK-3475) with a combination of MK-3475 (pembrolizumab) and BCG. All patients were evaluated for Grade 3 and higher adverse events considered related or possibly related to the addition of pembrolizumab to the treatment regimen. Due to the small sampling of subjects, no statistical analysis will be performed. Descriptive statistics in the form of counts calculated as percentages will be reported.
Measure: Count of Participants; unit: Participants
Groups:
- Intravenous MK-3475-100 mg/ Intravesical BCG: 3 subjects will be treated at a dose of 100 mg MK-3475 at 100 mg every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses
  Intravenous MK-3475/ Intravesical BCG: 6 cycles (each cycle is 21 days) of pembrolizumab will be given over 19 weeks in combination with BCG. BCG treatment will begin on Day 1 of cycle 3 of pembrolizumab.
Arm/Group | Intravenous MK-3475-100 mg/ Intravesical BCG | Intravenous MK-3475-200 mg/ Intravesical BCG
Number analyzed (Participants) | 3 | 10
Participants
  Number of Subjects with Grade 3, 4, or 5 treatment related adverse event(s) | 0 | 4
  Number of Subjects without a Grade 3, 4, or 5treatment related adverse event(s) | 3 | 6

2. Secondary Outcome: Number of Participants Without Bladder Tumors Upon Cystoscopy Following Treatment.
Description: Complete response rate per cystoscopy assessment of the bladder at 19 weeks from start of treatment with MK-3475 (pembrolizumab) at week 1.Subjects presenting at Week 19 with a bladder free of tumors upon cystoscopy and without local or metastatic spread were considered a complete response.. Suspicious lesions would be biopsied and sent for confirmation of pathology. Due to the small sampling of subjects, no statistical analysis will be performed. Descriptive statistics in the form of counts calculated as percentages will be reported.
Time Frame: 19 weeks
Population: Subjects presenting at Week 19 for cystoscopy with a bladder free of tumors or local or metastatic spread would be considered a complete response. Suspicious lesions would be biopsied and sent for confirmation of pathology.
Measure: Count of Participants; unit: Participants
Groups:
- Intravenous MK-3475-100 mg/ Intravesical BCG: 100 mg MK-3475 at 100 mg every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial (50mg) intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses starting at week 7.
- Intravenous MK-3475-200 mg/ Intravesical BCG: 200 mg MK-3475 at 100 mg every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial (50mg) intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses starting at week 7.
Arm/Group | Intravenous MK-3475-100 mg/ Intravesical BCG | Intravenous MK-3475-200 mg/ Intravesical BCG
Number analyzed (Participants) | 3 | 09
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: Each subject had adverse events collected from the time of consent through 30 days post-treatment completion with MK-3475/pembrolizumab. This was up to 23 weeks from the time of first treatment with MK-3475/pembrolizumab.
Groups:
- Intravenous MK-3475-100 mg/ Intravesical BCG: 3 subjects will be treated at a dose of 100 mg MK-3475 at 100 mg every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial (50mg) intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses
- Intravenous MK-3475-200 mg/ Intravesical BCG: Up to 12 subjects will be treated at a dose of 200 mg MK-3475 at 100 mg every 3 weeks (Q3W) intravenously (IV) for 6 doses and 1 vial (50 mg) intravesicular BCG suspended in 50 ml preservative-free saline once per week of 6 weekly doses
Arm/Group | Intravenous MK-3475-100 mg/ Intravesical BCG | Intravenous MK-3475-200 mg/ Intravesical BCG
All-Cause Mortality (participants affected / at risk) | 0/3 | 3/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 6/10
Other Adverse Events (participants affected / at risk) | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous MK-3475-100 mg/ Intravesical BCG (N=3) | Intravenous MK-3475-200 mg/ Intravesical BCG (N=10)
arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — arthritis of hands, shoulders, hips and knees
adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
thrombormbolic event (Vascular disorders) | 0 (0) | 1 (1) — pulmonary embolism
cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
neuropathy (Nervous system disorders) | 0 (0) | 1 (1) — motor neuropathy of lower right extremity
hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) — Asymptomatic hyperthyroidism defined by thyroid stimulating hormone and T4 levels.
injection site reaction (General disorders) | 0 (0) | 1 (2) — right hand redness and edema
pain-extremity (General disorders) | 0 (0) | 1 (1) — bilateral wrist pain
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
intra-operative hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) — secondary to cystoscopy discovery of friable tumor.
cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous MK-3475-100 mg/ Intravesical BCG (N=3) | Intravenous MK-3475-200 mg/ Intravesical BCG (N=10)
elevated Blood Urea Nitrogen (BUN) (Investigations) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
allergic rhinitis (General disorders) | 1 (1) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
anxiety (Nervous system disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
elevated AST (Investigations) | 0 (0) | 1 (1)
thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
chills (General disorders) | 0 (0) | 3 (3)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cystitis non-infective (Renal and urinary disorders) | 2 (3) | 6 (11)
darkening of hair (General disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
edema-limb (General disorders) | 1 (2) | 2 (2)
fatigue (General disorders) | 1 (1) | 8 (10)
fever (General disorders) | 0 (0) | 2 (2)
flu like symptoms (General disorders) | 0 (0) | 3 (5)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (1) | 3 (5)
jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypersomnia (General disorders) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) — bladder
injection site reaction (General disorders) | 0 (0) | 1 (1) — IV site infiltrated
insomnia (General disorders) | 2 (2) | 3 (3)
increased protein in urine (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
axonal neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
ocular redness (Eye disorders) | 0 (0) | 1 (1)
otitis externa (Infections and infestations) | 0 (0) | 1 (1)
toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
intestinal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
prostatic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
sinusitis (Infections and infestations) | 1 (1) | 0 (0)
paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
weight loss (Investigations) | 0 (0) | 1 (1)
Elevated leukocytes in urine (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study is limited by the small number of subjects treated and evaluated which did allow for statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT02324582/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT02324582/ICF_001.pdf